CLINICAL TRIAL: NCT05510206
Title: The Effectiveness of SmartArch Versus Super Elastic Nickel-titanium Aligning Archwires: a Randomized Clinical Trial
Brief Title: SmartArch vs Super Elastic NiTi Aligning Archwires
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Omar Khairullah Ahmed, Orthodontics master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 611422
Record Dates: First submitted 2022-08-02; First posted 2022-08-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: lower anterior crowding

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super elastic NiTi Group (Active Comparator): 0.014-inch super elastic nickel-titanium archwire (ortho Technology™ , west Columbia, USA) will be placed in mandibular arch at the day of bonding. Eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks.
  Interventions: Device: Leveling and alignment
- Smartarch Group (Experimental): 0.016-inch Smartarch archwir (Ormco™, USA) will be placed in mandibular arch at the day of bonding. Re-ligated every four weeks for 16 weeks.
  Interventions: Device: Leveling and alignment

INTERVENTIONS:
Device: Leveling and alignment — Polishing, Bonding of appliance, placement of the first arch wire for Super elastic NiTi group then the second wire after two months taking study model each month during the study For Smartarch Group placing experimental arch wire for 4 months , taking impression each month.
  For both groups peri-apical X-Ray to lower anterior teeth is taken prior to treatment and 4 months later, also visual pain analogue scale is taken for 7 days after placing archwires

SUMMARY:
This study is intended primarily to compare the alignment efficiency and rate of two different types of archwires that are used in the first stage of orthodontic treatment , also addressing pain and root resorption that may be associated during treatment, with the hypothesis being a consideration of no deference between the two archwires.

DETAILED DESCRIPTION:
This will be a multicenter non-stratified prospective randomized clinical trial with parallel groups trial with equal randomization (1:1 allocation ratio), two public orthodontic center will allocate patients for this trial. The patients will be initially assessed for eligibility to be included in the study by the investigator. Those who will meet the inclusion criteria will be informed about the nature of the study verbally to take the initial approval for participation. Then they will be provided by the patient information sheet and consent form, which explains the nature of the study, to read carefully at home and provide their decision about participation at the subsequent appointment. If the patient age below 18 years, parent assent should be taken. Any further enquiries regarding the study by the patient should be resolved by the investigator on the second visit.

The patients will be treated with straight wire appliance using MBT prescription brackets with 0.022-inch slot (Pinnacle®, Ortho Technology, USA). Bracket placement will be standardized using a height gauge. Initially, teeth polishing will be performed with pumice and rubber cup for 10 seconds using a low-speed handpiece, followed by water rinsing and air drying (oil-free air spray for 30 seconds). Bonding technique will be standardized as follows:

* Teeth etching with 37% phosphoric acid gel for 30 seconds.
* Rinsing thoroughly (5 seconds per tooth for liquid etchant and 10 seconds per tooth for gel etchant) to stop the etching process and to remove demineralized particles then air drying until the white frosty appearance of the etched surface is observed.
* Application of a thin layer of Light Bond™ Sealant (Reliance®, Itasca, USA) for one minute and air application for 5 seconds.
* Bonding of brackets and tubes using Light Bond™ light cure orthodontic adhesive (Reliance®, Itasca, USA) applied on their bases and light-cured above interproximal contacts at a distance of 2-3 mm (5 seconds mesially and 5 seconds distally for brackets and 10 seconds mesially and 10 seconds occlusally for molar tubes).

All the participants will receive a standardized treatment protocol. At the day of bonding, 0.016-inch archwire will be placed for the Smartarch group. It will be re-ligated every four weeks. While, for the super elastic NiTi group, 0.014-inch archwire will be placed at the day of bonding and eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks. Archwires will be tied to the bracket by elastomeric modules, with laceback of canines to first molars. If there is any debonding during treatment, this should be dealt with as an emergency case and re-bonded within 24 hours, otherwise the case will be considered as dropout. Since this study will be performed during the initial phase of treatment, no deviation in the protocol of treatment will be accepted (such as adding additional archwire in the sequence or using power chain). A good-quality alginate impression for the lower arch should be taken pre-treatment and after 4, 8, 12 and 16 weeks and a stone study model is obtained. Periapical X-ray for the mandibular central incisors will be taken pre-treatment and after 16 weeks. The participants will be provided by a visual analog scale (0-10) to record their pain perception during the first week after each wire placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for fixed appliance orthodontic treatment with 5-9 mm crowding of mandibular anterior teeth according to Little's irregularity index (LII).
* Presence of all mandibular permanent teeth, except the third molars.
* Overbite and overjet that do not interfere with bracket placement on mandibular anterior teeth.
* No history of trauma or root resorption in the mandibular incisors.

Exclusion Criteria:

* Previous orthodontic treatment.
* Less than 5mm of mandibular incisor crowding (LII).
* Blocked-out teeth that cannot be engaged with the aligning archwire.
* Prior experience of periodontal disease and loss of attachment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Changes in alignment of anterior teeth will be measured using Little's irregularity index | 16 weeks
  A good-quality alginate impression for the lower arch should be taken pre-treatment and after 4, 8, 12 and 16 weeks and a stone study model is obtained. This study model which should be free from any discrepancy (such as bubbles) will be used to measure Little's irregularity index using a digital Vernier caliper to calculate the amount of mesial and distal contact displacement from the mesial contact surface of right mandibular canine to that on the other side, to the nearest 0.01 mm. The sum of these measurements represents the amount of Little's irregularity index.

SECONDARY OUTCOMES:
Root resorption incidence using the scoring index that was provided by Malmgren et al. (1982) | 16 weeks
  assessed by scoring system for orthodontic induced apical root resorption from (0-3) on Root resorption will be evaluated for the mandibular central incisors using periapical radiographs with digital sensors, and the worst score for either left or right central will be taken using the scoring index by Malmgren et al. (1982):
  Grade 1: Irregular apical root contour. Grade 2: Minor apical root resorption, a small area of root loss amounting to less than 2 mm.
  Grade 3: Severe apical root resorption from 2 mm to one third of the original root length.
  Grade 4: Extreme apical root resorption exceeding one third of the original root length.
Pain perception using visual analog scale | 1st week after wire placement
  Evaluations of pain/discomfort will be made in the evening on a daily basis over the first seven days after bonding using a 10-point visual analog scale (VAS) with 0 refers to "no pain" and 10 refers to "intolerable pain". The participants will be reminded daily by a phone call or a text message to mark the recording sheet and will be asked to bring it on their next appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Ammar S. Kadhum, Asst. Prof., Study Director — University of Baghdad
Locations (1):
- University of Baghdad\ College of Dentistry, Baghdad, Bab Al-Moadham, Iraq

IPD SHARING:
Plan to Share IPD: Yes
It will be available on request.

REFERENCES:
- [Background] Malmgren O, Goldson L, Hill C, Orwin A, Petrini L, Lundberg M. Root resorption after orthodontic treatment of traumatized teeth. Am J Orthod. 1982 Dec;82(6):487-91. doi: 10.1016/0002-9416(82)90317-7. PMID 6961819
- [Background] Nabbat SA, Yassir YA. A clinical comparison of the effectiveness of two types of orthodontic aligning archwire materials: a multicentre randomized clinical trial. Eur J Orthod. 2020 Dec 2;42(6):626-634. doi: 10.1093/ejo/cjz102. PMID 32011678
- [Background] Wang Y, Liu C, Jian F, McIntyre GT, Millett DT, Hickman J, Lai W. Initial arch wires used in orthodontic treatment with fixed appliances. Cochrane Database Syst Rev. 2018 Jul 31;7(7):CD007859. doi: 10.1002/14651858.CD007859.pub4. PMID 30064155
- [Derived] Noori RM, Ahmed OK, Kadhum AS, Yassir YA, Di Blasio M, Russo D, Cicciu M, Minervini G. The Effectiveness of Conventional and Advanced Aligning Archwires: The Insights of Two Randomized Clinical Trials. Eur J Dent. 2025 Oct;19(4):985-997. doi: 10.1055/s-0044-1795080. Epub 2025 Apr 4. PMID 40185146